CLINICAL TRIAL: NCT02062944
Title: Liver Transplant Tolerance Enhanced By Sirolimus Therapy
Brief Title: SRL (Sirolimus) Withdrawal
Acronym: SRL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Josh Levitsky, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00072766
Record Dates: First submitted 2014-02-03; First posted 2014-02-14 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Acute Rejection of Liver Transplant; Effects of Immunosuppressant Therapy
Keywords: Liver Transplant; Sirolimus; Rapamune; Immunosuppressant Therapy; Withdrawal
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm study Sirolimus Withdrawal (Experimental): SRL minimization will be performed if clinically, biochemically and histologically stable. Patients entering the minimization phases will be reduced every month by 50% of total dose of Sirolimus until they reach .5mg daily for one month. Then .5 mg every other day, then twice weekly, the once weekly dosing. This should take approximately 6 month to complete minimization. Liver function tests will be monitored every 2 weeks. For any patient developing liver dysfunction, liver biopsy will be performed. Patients will then be completely withdrawn and followed post-withdrawal for 12 months.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — SRL minimization will be performed if clinically, biochemically and histologically stable. Patients entering the minimization phases will be reduced every month by 50% of total dose of Sirolimus until they reach .5mg daily for one month. Then .5 mg every other day, then twice weekly, the once weekly dosing. This should take approximately 6 month to complete minimization. Liver function tests will be monitored every 2 weeks. For any patient developing liver dysfunction, liver biopsy will be performed. Patients will then be completely withdrawn and followed post-withdrawal for 12 months.
  Other Names: Withdrawal from Immunosuppressant Therapy; Minimization of Immunosuppressant Therapy

SUMMARY:
The significance of this clinical trial lies in its potential to increase the success of immunosuppression (IS) therapy withdrawal in liver transplant (LT) recipients, thus decreasing the negative impact of IS on their long-term outcomes. Lifetime immunosuppression (IS) with standard agents, the calcineurin inhibitors (CNI) cyclosporine and tacrolimus (TAC), is currently required at clinically recommended doses and trough levels to prevent allograft rejection. However, this occurs at the significant expense of long-term CNI toxicity, i.e. chronic kidney disease (CKD), hypertension, hyperlipidemia, diabetes, infections and malignancy. With improvements in early graft and patient survival, long term adverse IS effects have become increasingly important in this rapidly expanding patient population. The strategies to reduce long term CNI toxicity include dose minimization that still leaves patients on CNI therapy, conversion to non-CNI therapy, or even complete IS withdrawal. The second approach, conversion to non-CNI IS therapy, is attractive in the potential to stabilize or improve renal function and other CNI toxicities. One such non-nephrotoxic IS agent, the mammalian target of rapamycin inhibitor (mTOR-I) SRL, has a different mechanism of IS action and studies have shown that CNI to SRL conversion can stabilize renal dysfunction with a low risk of rejection. Yet even with these possible benefits, patients on SRL are still subject to lifetime IS therapy with side effects and costs, highlighting the need to investigate the strategies that promote full IS withdrawal without rejection (3rd approach), also known as 'operational tolerance'.

DETAILED DESCRIPTION:
Study Overview The study proposed is a prospective trial of controlled SRL monotherapy minimization and withdrawal in up to 25 stable non-immune non-viremic LT recipients. Given the sample size calculations (see Statistical section), we plan to enroll up to 25 SRL monotherapy patients for this study (Figure 1). All patients will be consented to undergo laboratory evaluation as well as an enrollment liver biopsy and blood tests. If the patient meets inclusion/exclusion (I/E) criteria (see below), SRL will be minimized over 6 months until once a week dosing is achieved. Repeat clinical and immunological blood tests as above will be performed, and if no biochemical signs of rejection, SRL will be discontinued with blood tests and liver biopsy 12 months later for similar biochemical, histological and immunological measures. At any concern for rejection, liver biopsy and assays for equivalent biochemical, histological and immunological measures will be performed and if rejection is diagnosed on biopsy, a second attempt at withdrawal will not be performed. Patients will be monitored as standard of care with clinic visits every 6 months and laboratory tests every 2 weeks. The total study length will be 18 months: 6 month minimization phase and 1 year follow-up after withdrawal success/failure. The primary outcome will be the proportion of tolerant patients off SRL therapy with normal liver biochemistry and graft histology at 18 months. Secondary outcomes will include the incidence, severity and reversibility of rejection, patient/graft survival, resolution of SRL and other non-specific IS effects, and the assessment of clinical/immunological biomarkers of tolerance. All continuous/categorical clinical variables will be compared with the appropriate statistical analyses.The goal is that the primary and secondary aims will provide valuable preliminary data to further elucidate the mechanisms of mTOR-I immunoregulation and for determining the initial clinical success/feasibility of the mTOR-I approach (vs. historical 20% CNI withdrawal success seen in studies from the Immune Tolerance Network [ITN] and other groups). This is all so as to guide a submission to the Immune Tolerance Network for larger, more adequately powered prospective trials comparing SRL vs. CNI withdrawal and accompanying biomarker predictors of tolerance. If this pilot study fails to show a correlation between our biomarkers and the success/failure of SRL withdrawal, or is associated with an unacceptable low (e.g. <20%) rate of operational tolerance, then this would avoid the necessity for such large, expensive trials and support the continued development of alternative approaches to tolerance.

Consent and Initial Phase of Enrollment (see Study Protocol Figure- Appendix A) These liver transplant candidates (up to 25 SRL) will be approached for consideration and informed consent into the study. The consent form will include discussion of the risks/benefits of their current therapy (SRL) and the planned minimization/withdrawal. Specifically, the risks of minimization/withdrawal (i.e. developing acute or chronic rejection, alloimmune hepatitis during any portion of the study), although unlikely, will be a major emphasis of the consent process. The consent form will also include the strict requirement for patients to follow all instructions from the PI in regard to the close laboratory follow-up occurring throughout the trial, to diagnose any episode of rejection or concern as early as possible to be able to respond appropriately. All of the study procedures will be discussed with the patient during clinic visits. They will be informed that neither participation nor refusal will influence their clinical care. All laboratory tests or costs related to their care in the study, with the exception of non-standard of care items (i.e. liver biopsies, blood assays), will be the responsibility of the patient and/or his/her insurance company. They will be asked questions afterwards to verify comprehension and then sign the consent form documenting their agreement to participate. A signed copy of the consent form will be given to them. Participation is completely voluntary and they may discontinue participation the study at any time without affecting their care or participation in any other study. No financial compensation will be given.

Screening Evaluation at Enrollment (see Study Protocol Figure) After long term (> 3 years post-LT, > 3 months on SRL monotherapy) on SRL monotherapy, inclusion/exclusion criteria will be reviewed and if appropriate, consent as above will be obtained. If the patient agrees and signs consent, baseline standard of care screening laboratories complete blood count, comprehensive metabolic panel, sirolimus (CBC, CMP, SRL trough level, fasting lipid profile, hemoglobin A1C [HbA1C], urine protein/creatinine ratio) and non-standard of care biomarker assays (blood immunophenotyping, proteogenomics) and liver biopsy (histology and graft immunohistochemistry) will be performed as dictated by the protocol. In addition, the liver biopsy will be used to determine stability in graft function (i.e. no evidence of rejection or immune-mediated hepatitis) before considering minimization/withdrawal. SRL minimization/withdrawal will only be performed if clinically, biochemically and histologically [by biopsy; liver transplant pathology read (Yang, Rao)] stable. Throughout the entire study, liver function tests will be monitored every 2 weeks (monthly is standard of care, so the interim non-standard of care 2 week blood tests will be covered by the study funds). Patients entering the minimization/withdrawal phases will be reduced by a total dose of 50% of their baseline dose every month until patients are on 0.5 mg SRL daily. At this point, every other day dosing will begin x 1 month. If no LFT abnormalities, twice weekly dosing x 1 month, then once a week dosing x 1 month. Prior to complete discontinuation, repeat clinical (screening labs above) and blood biomarker assays (blood immunophenotyping, proteogenomics) will be performed. Liver biopsy will not be performed at this juncture unless there are biochemical signs of liver injury. If complete withdrawal is deemed safe (no evidence of biochemical abnormalities) patients will be withdrawn completely (i.e. the once/week SRL dose discontinued) and followed off IS therapy for one year. In this time period, liver function tests will be monitored every 2 weeks, as usual, and repeat clinical (screening labs above), liver biopsy and blood (blood immunophenotyping, proteogenomics) assays performed at the end of this year or at any concern for rejection.

Blood and Tissue Samples Standard of care laboratories (CBC, CMP) will be performed every month on all patients, and only LFTs performed in the interim 2 weeks between each month (non-standard of care; covered by the study funds) until complete withdrawal. 3 green top 5 mL and 3 red top 5 mL tubes of blood for biomarker assays will be taken on all patients prior to study enrollment, prior to complete withdrawal, and one year after withdrawal or at the time of suspected rejection. Liver biopsy (one 3 cm biopsy- 2 cm for histology and 1 cm for genomic assays) will be performed at baseline (pre-minimization) and 1 year post withdrawal. A separate clinical informed consent will be obtained each time a liver biopsy is performed. If the patient develops elevation in liver transaminases requiring a liver biopsy at any stage of the study protocol, blood (all for immune monitoring (IM) assays) will be requested from the patient at the time of the biopsy. If rejection occurs, the patient will be followed in the study until completion but not be further withdrawn from SRL or have a liver biopsy at the end of the study

Follow-up Laboratory follow-up is described above- every 2 weeks throughout the trial until complete withdrawal. Any biochemical (or clinical) signs or significant liver function test abnormalities will be acted on immediately either by liver biopsy or a pause in IS withdrawal per investigator discretion. All patients will be seen in the clinic every 3 months to assess for any new signs or symptoms or resolution of drug side effects in the minimization or withdrawal arm. Quality of life questionnaires; Post Liver Transplant Quality of Life Instrument (pLTQ) and the Promis-29 profile v1.0 will be administered at the study onset and after successful vs. unsuccessful withdrawal (end of study)

Outcome Measures The primary outcome will be the proportion of patients off SRL therapy with normal liver biochemistry and graft histology at 12 months (i.e. tolerant). Thus, the incidence of graft dysfunction (acute rejection, immune mediated or autoimmune hepatitis, chronic rejection) or non-tolerance will be assessed in this SRL withdrawal group and compared to the historical CNI group (20% tolerant; 80% failure) as the primary endpoint. This rate will be a composite of the cumulative number of biopsy-proven graft dysfunctions requiring conversion back to SRL or additional IS therapy or discontinuation of minimization/withdrawal that occur during the course of the study. Major secondary measures compared will be the predictive capacity of the blood and graft biomarker assays (immunophenotyping, genomic/proteomics) before and after minimization/withdrawal in the success vs. failure groups. Clinical secondary outcomes will be compared: the number of infectious complications, liver biopsy complications, cardiovascular outcomes (i.e. blood pressure, diabetes control, lipid levels), renal function, hematopoietic parameters, gastrointestinal effects, or other side effects of SRL that may or may not improve or develop with minimization/withdrawal. These will all be documented by a study database during patient visits, electronic charts and/or by phone communication. Finally, quality of life (Post Liver Transplant Quality of Life Instrument (pLTQ) and the Promis-29 profile v1.0) will be analyzed at the end of the study to determine the effect of IS minimization/withdrawal on other health benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female recipients of all races, ≥ 18-75 years of age
2. Patients who underwent primary living or deceased donor liver transplantation ≥ 3 years (previous to screening ) and on ≥ 3 months of stable SRL monotherapy
3. Recipient of single organ transplant only
4. Liver transplant for non-immune, non-viral (no hepatitis B or hepatitis C virus unless currently non-viremic) causes
5. Ability to provide informed consent and to comply with the study protocol of IS withdrawal.

Exclusion Criteria:

1. Inability or unwillingness to provide informed consent
2. Acute cellular rejection within 12 months prior to enrollment
3. Viral (viremic hepatitis B virus [HBV] or hepatitis C virus [HCV]) or immune-mediated liver disease (Autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cirrhosis) history
4. Abnormal liver function tests: Direct bilirubin ≥ 1 mg/dL; ([ALT, AST, GGT] or alkaline phosphatase [AlkPhos] ≥ 2x [ULN]); 5) Abnormal graft histology at enrollment: a) ≥ Grade 2 inflammation or stage 2 fibrosis; b) Acute or Chronic Rejection; c) De-novo Autoimmune Hepatitis; d) inflammation of >50% of portal tracts; e) Other pathology not-specified but deemed high risk per the PI and pathologist; 6) Ongoing or recurrent substance abuse

7) Retransplantation or combined liver-other organ 8) Human Immunodeficiency Virus(HIV) co-infection 9) Glomerular Filtration Rate (GFR)<30 ml/min by estimated glomerular filtration rate ([eGFR]-[MDRD-4])

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Levitsky J, Burrell BE, Kanaparthi S, Turka LA, Kurian S, Sanchez-Fueyo A, Lozano JJ, Demetris A, Lesniak A, Kirk AD, Stempora L, Yang GY, Mathew JM. Immunosuppression Withdrawal in Liver Transplant Recipients on Sirolimus. Hepatology. 2020 Aug;72(2):569-583. doi: 10.1002/hep.31036. Epub 2020 Jun 8. PMID 31721246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To identify our cohort, we screened our database for all living LTRs transplanted at Northwestern (1995-2012) who met the following inclusion criteria: (1) adult LTR ≥18 years of age, (2) ≥3 months of SRL monotherapy with trough levels of 3-8 ng/mL, and (3) ≥3 years post-LT (primary living or deceased donor).
Pre-assignment Details: Baseline physical examination and laboratory tests were performed, and if acceptable per the criteria above, a baseline liver biopsy was performed within 1 month. Patients were excluded from IS withdrawal if any of the following were present on local biopsy read: (1) ≥grade 2 inflammation or stage 2 fibrosis, (2) acute or chronic rejection, (3) de novo autoimmune hepatitis, (4) inflammation of > 50% of portal tracts, and (5) other pathology not specified but deemed high risk per the pathologist.
Period: Overall Study
Arm/Group | Single-arm Study Sirolimus Withdrawal
Started | 21
Completed | 15
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — New hemotological disorder identified | 1
Not completed — Uncontrolled Hypertension | 1
Not completed — underwent pre-weaning biospsy and excluded for mild subclinical ACR | 3

BASELINE CHARACTERISTICS:
Arm/Group | Single-arm Study Sirolimus Withdrawal
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Tolerant Patients Off SRL Therapy With Normal Liver Biochemistry and Graft Histology at 12 Months
Description: The primary outcome will be the proportion of patients off SRL therapy with normal liver biochemistry and graft histology at 12 months (i.e. tolerant). Thus, the incidence of graft dysfunction (acute rejection, immune mediated or autoimmune hepatitis, chronic rejection) or non-tolerance will be assessed in this SRL withdrawal group and compared to the historical CNI group (20% tolerant; 80% failure) as the primary endpoint.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm Study Sirolimus Withdrawal
Number analyzed (Participants) | 15
Participants | 8

2. Secondary Outcome: Number of Subjects With TCMR Rejection
Description: Major secondary measures compared will be the predictive capacity of the blood and graft biomarker assays (immunophenotyping, genomic/proteomics) before and after minimization/withdrawal in the success vs. failure groups.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm Study Sirolimus Withdrawal
Number analyzed (Participants) | 15
Participants | 6

3. Other Pre Specified Outcome: Number of Participants Resumed SRL After Minimization
Description: patient did not have rejection during withdrawal but was withdrawn from the trial due to an unexpected adrenal metastasis of hepatocellular carcinoma.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm Study Sirolimus Withdrawal
Number analyzed (Participants) | 15
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Single-arm Study Sirolimus Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm Study Sirolimus Withdrawal (N=15)
biopsy-proven mild rejection (Hepatobiliary disorders) | 1 (1) — Patient had abdominal pain, hospitalized, emergency CT scan showed adhesions. Patient discharged on 4th day. Subject taken off study 1 month prior due to a biopsy-proven mild rejection and started on IS and monitored.
Stool in blood after biopsy (Hepatobiliary disorders) | 1 (1) — Subject seen for a study specific biopsy and after returning home had two episodes of watery stool with blood in stool. Patient instructed to go to emergency room if another episode. The following day bleeding less vitals normal. No further bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT02062944/Prot_SAP_000.pdf